CLINICAL TRIAL: NCT00508144
Title: Single Agent Alimta in Poor Performance Status in Patients With Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Single Agent Alimta in Poor Performance Status in Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-0957; NCI-2012-01581 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2007-07-26; First posted 2007-07-27 (Estimated); Results first posted 2017-02-13 (Actual); Last update posted 2017-02-13 (Actual); Status verified 2016-12

CONDITIONS: Lung Cancer
Keywords: Non-Small Cell Lung Cancer; Lung Cancer; NSCLC; Malignant pleural effusion; Pericardial effusion; Pemetrexed; Alimta; LY231514; Poor Performance Status; Asymptomatic Brain Metastases
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Pleural Effusion, Malignant; Pericardial Effusion | interventions — Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Alimta (Experimental): Alimta 500 mg/m^2 by vein Once Over 10 Minutes Every 3 Weeks.
  Interventions: Drug: Alimta

INTERVENTIONS:
Drug: Alimta — 500 mg/m^2 by vein Once Over 10 Minutes Every 3 Weeks
  Other Names: Pemetrexed; LY231514; MTA; Multitargeted Antifolate; NSC-698037

SUMMARY:
The goal of this clinical research study is to learn how effective the drug pemetrexed (ALIMTA®) is in treating advanced NSCLC in patients with poor performance status (PS) (inability to perform every day activities without difficulty).

Objectives:

Primary Objectives:

* PS = 2 cohort: Response
* PS = 3 cohort: Descriptive

Secondary Objectives:

* Tolerability of single agent pemetrexed (Alimta®) in PS = 3 NSCLC patients
* Improved symptoms (both cohorts)
* Molecular Correlative studies (both cohorts)
* Overall survival
* Time to progression

DETAILED DESCRIPTION:
Pemetrexed is designed to block enzymes in the body that are important for tumor growth. Pemetrexed is commercially approved for the treatment of NSCLC but not for poor performance status patients.

If participants are found to be eligible to take part in this study, they will receive pemetrexed once every 3 weeks through a needle in their vein over about 10 minutes. Every 3 weeks is considered 1 treatment cycle. Once the treatment has started, they will return to the clinic before every treatment cycle. At these visits, they will have a physical exam, a performance status evaluation, and routine blood (about 3-4 teaspoons) and urine tests. They will have a chest x-ray and will be asked to complete a questionnaire about how you are feeling. they will also have a CT or MRI scan after Cycle 1 and every odd cycle from then on.

They are required to take folic acid by mouth every day for 5 days before the first dose of pemetrexed and continuing until 3 weeks after your last dose of pemetrexed. They will also receive an injection of vitamin B12 into your muscle before first dose of pemetrexed. The vitamin B12 injection will be repeated every 9 weeks until 3 weeks after their last dose of pemetrexed.

They will also to take a few low-dose steroid (dexamethasone) tablets twice a day before treatment, the day of treatment, and the day after each treatment. These will be taken to decrease the risk of rash and nausea caused by pemetrexed.

They may continue treatment with pemetrexed until your tumor grows or an unacceptable side effect occurs. They will be evaluated for symptoms 1-2 times per week while you are receiving treatment and then 2 weeks after stopping study treatment until 6 months after stopping treatment.

When they stop treatment on this study, they will have a physical exam, routine blood (3-4 teaspoons) and urine tests, and a chest x-ray. The study doctor may ask them to visit University of Texas MD Anderson Cancer Center or be contacted by phone for follow-up on how they are doing.

This is an investigational study. The FDA has approved pemetrexed for the treatment of advanced NSCLC after earlier treatment with chemotherapy, and for the treatment for malignant mesothelioma in combination with cisplatin. About 70 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically proven Stage IIIB (T4 lesion due to malignant pleural or pericardial effusion) or Stage IV. Clinically significant pleural or peritoneal effusions should be drained prior to dosing.
2. Zubrod PS 2 or PS 3
3. Patients with asymptomatic brain metastases and no requirement for corticosteroids or anticonvulsants are eligible for this clinical trial.
4. Measurable OR non-measurable disease documented by CT or MRI.
5. Patients may have had </=1 prior chemotherapy regimens but multiple prior biologic regimens. At least 4 weeks need to have elapsed since last chemotherapy or biologic therapy administration.
6. Prior radiation therapy is permitted; however, at least two weeks must have elapsed since the completion of prior radiation therapy and patients must have recovered from all associated toxicities at the time of registration. Measurable or non-measurable disease must be outside the previous radiation field OR patients with visible progression or new lesions within the radiation field are eligible.
7. At least two weeks must have elapsed since surgery and patients must have recovered from all associated toxicities at the time of registration.
8. Creatinine clearance >/= 45 cc/min measured or calculated using the following formula: Calculated Creatinine Clearance = (140 - age) X WT (kg) X (0.85 if female)/72 X creatinine (mg/dl) Calculated Creatinine Clearance = (140 - age) X WT (kg) X (1.00 if male)/72 X creatinine (mg/dl)
9. Absolute neutrophil count (ANC) >/= 1,500/µl
10. Platelet >/= 100,000/µl
11. ALT/AST: </=3.0 x upper limit of normal (ULN) except in known hepatic metastasis wherein may be </= 5 x ULN
12. Bilirubin: </=1.5 x ULN
13. Hemoglobin: >/=9.0 x 10^9/L
14. Patient must not be pregnant or breastfeeding. Patients of childbearing potential agree to practice an effective contraceptive method for the duration of the study.
15. Patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines.
16. Men and women, aged >/=18 years.

Exclusion Criteria:

1. Prior treatment with pemetrexed therapy.
2. Patients planning to receive any other concomitant anticancer treatment including chemotherapy, radiation therapy, biologic agents or any other investigational drugs.
3. Women who are pregnant or breastfeeding may not participate in this trial. All women of childbearing potential must have a negative pregnancy test within 24 hours prior to enrolling in the study.
4. Inability to interrupt aspirin or other nonsteroidal anti-inflammatory agents for a 5-day period (8-day period for long-acting agents, such as piroxicam).
5. Inability and unwillingness to take folic acid or vitamin B12 supplementation.
6. Inability to take corticosteroids.
7. Prior malignancy except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated Stage I or II cancer from which the patient is currently in complete remission or other cancer from which the patient has been disease-free for >/= 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2005-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Zinner, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: September 1, 2005 to June 30, 2011. All recruitment done at The University of Texas MD Anderson Cancer Center.
Pre-assignment Details: Of the 64 participants registered, fifty-eight (58) were eligible, four (4) were invaluable, and six (6) were not eligible to participate in this trial.
Period: Overall Study
Arm/Group | Alimta
Started | 64
Completed | 53
Not Completed | 11
Not completed — Not eligible | 6
Not completed — Death | 5

BASELINE CHARACTERISTICS:
Arm/Group | Alimta
Number analyzed (Participants) | 64
Age, Continuous [Median (Full Range); unit: years] | 68 [45 to 88]
Gender [Count of Participants; unit: Participants]
  Female | 24
  Male | 40
Region of Enrollment [Number; unit: participants]
  United States | 64

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (OR) Where OR=CR+PR: Number of Participants With Responses of Complete Response (CR) and Partial Response (PR)
Description: Complete Response (CR): Complete disappearance of all measurable & non-measurable disease; No new lesions; No disease related symptoms; Normalization of markers & other abnormal lab values.
  Partial Response (PR): Applies only to those with at least one measurable lesion. >/= 30% decrease under baseline of sum of longest diameters of all target measurable lesions. No unequivocal progression of non-measurable disease. No new lesions. All target measurable lesions assessed using same techniques as baseline.
  Progression: 20% increase in sum of longest diameters of target measurable lesions over smallest sum observed (over baseline if no decrease during therapy) using same techniques as baseline. Unequivocal progression of non-measurable disease in opinion of treating physician.
  Evaluated for symptoms 1-2 times per week while receiving treatment then 2 weeks after stopping study treatment (expected 4 cycles).
Time Frame: Evaluated with 3 week treatment cycles, up to 4 cycles or 12 weeks
Population: Of 58 eligible participants, only 54 treated were available for response and five (5) experienced an early death, five (5) were later deemed inevaluable, and two had an indeterminate response.
Measure: Count of Participants; unit: Participants
Arm/Group | Alimta
Number analyzed (Participants) | 42
Participants | 3

ADVERSE EVENTS:
Time Frame: Adverse event data collected for three-week treatment cycle, up to four cycles or 12 weeks.
Arm/Group | Alimta
Serious Adverse Events (participants affected / at risk) | 32/58
Other Adverse Events (participants affected / at risk) | 43/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alimta (N=58)
Death (General disorders) | 5 (5)
ANEMIA (Blood and lymphatic system disorders) | 6 (6)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1)
BRONCHIECTASIS EXACERBATION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
BRONCHITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
CARDIOPULMONARY ARREST (Cardiac disorders) | 1 (1)
CELLULITIS (Skin and subcutaneous tissue disorders) | 2 (2)
Chest Pain (General disorders) | 1 (1)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (COPD) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 3 (3)
HEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 3 (3)
HYPOTENSION (Vascular disorders) | 2 (2)
ISCHEMIC ILEITIS/COLITIS (Gastrointestinal disorders) | 1 (1)
LEFT FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 1 (1)
LEUKOPENIA (Blood and lymphatic system disorders) | 1 (1)
NEUTROPENIC FEVER (Blood and lymphatic system disorders) | 3 (3)
NONSUSTAINED VENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 (1)
PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 8 (8)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 2 (2)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
SEPTIC SHOCK (Infections and infestations) | 1 (1)
SINUS TACHYCARDIA (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alimta (N=58)
Alkaline phosphatase increased (Investigations) | 1 (1)
Alanine aminotransferase decreased (Investigations) | 2 (2)
Alanine aminotransferase increased (Investigations) | 2 (2)
ANEMIA (Blood and lymphatic system disorders) | 4 (4)
ANOREXIA (Metabolism and nutrition disorders) | 5 (5)
Aspartate aminotransferase increased (Investigations) | 5 (5)
ATRIAL FIBRILLATION (Cardiac disorders) | 2 (2)
Blood bilirubin increased (Investigations) | 1 (1)
BRONCHITIS (Infections and infestations) | 3 (3)
CANDIDIASIS (Reproductive system and breast disorders) | 1 (1)
CARDIOVASCULAR GENERAL (Cardiac disorders) | 1 (1)
COLITIS (Infections and infestations) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 2 (2)
CONSTITUTIONAL SYMPTOMS, FATIGUE (General disorders) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Creatinine increased (Investigations) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1)
DIARRHEA (Gastrointestinal disorders) | 1 (1)
DIZZINESS (Nervous system disorders) | 2 (2)
DRY MOUTH (Gastrointestinal disorders) | 2 (2)
DRY SKIN (Skin and subcutaneous tissue disorders) | 2 (2)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 8 (8)
EDEMA (General disorders) | 2 (2)
FATIGUE (General disorders) | 10 (10)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1)
FEVER NEUTROPENIC (Blood and lymphatic system disorders) | 3 (3)
FEVER UNKNOWN ORIGIN (General disorders) | 7 (7)
FEVER WITHOUT NEUTROPENIA (General disorders) | 2 (2)
GASTROINTESTINAL DISORDERS (Belly pain) (Gastrointestinal disorders) | 1 (1)
GLUCOSE, SERUM-HIGH (Metabolism and nutrition disorders) | 1 (1)
Hemoglobin increased (Investigations) | 16 (16)
HEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 3 (3)
HEMORRHAGE, PULMONARY (Respiratory, thoracic and mediastinal disorders) | 2 (2)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 2 (2)
HYPERKALEMIA (Metabolism and nutrition disorders) | 2 (2)
HYPERURICEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOGLYCEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOKALEMIA (Metabolism and nutrition disorders) | 6 (6)
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPONATREMIA (Metabolism and nutrition disorders) | 5 (5)
HYPOPHOSPHATEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOTENSION (Vascular disorders) | 1 (1)
INFECTION (Infections and infestations) | 3 (3)
INFECTION (OTHER) (Infections and infestations) | 1 (1)
INFECTION UNKNOWN (Infections and infestations) | 1 (1)
Infection with Normal White Blood Count (Infections and infestations) | 2 (2)
Infection with Normal Absolute Neutrophil Count (ANC) (Infections and infestations) | 5 (5) — Lung-pneumonia
INSOMNIA (Psychiatric disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2)
LYMPHOPENIA (Blood and lymphatic system disorders) | 2 (2)
MUCOSITIS (CLINICAL) (Gastrointestinal disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 9 (9)
Neutrophil count decreased (Investigations) | 3 (3)
Platelet count decreased (Investigations) | 5 (5)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 3 (3)
PULMONARY (OTHER) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RASH/DESQUAMATION (Skin and subcutaneous tissue disorders) | 3 (3)
RENAL/GENITOURINARY DISORDER (Renal and urinary disorders) | 1 (1)
SENSORY ALTERATION (Nervous system disorders) | 1 (1)
SINUS TACHYCARDIA (Cardiac disorders) | 1 (1)
STOMATITIS (Gastrointestinal disorders) | 1 (1)
SWEATING (Skin and subcutaneous tissue disorders) | 1 (1)
URINARY RETENTION (Renal and urinary disorders) | 1 (1)
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1)
WEIGHT LOSS (Investigations) | 3 (3)
WOUND INFECTION (Infections and infestations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes